CLINICAL TRIAL: NCT03861832
Title: A Systematic Medical Approach to Reward Transformation (SMART) for Brain Health in Opioid Use Disorder
Brief Title: SMART Brain Health in African-Americans
Acronym: SMART
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Howard University (Other)
Collaborators: Medical Home Development Group (Unknown); Geneus Health (Unknown)
Responsible Party: Principal Investigator, Marjorie Gondre-Lewis, Professor, Howard University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R41MD012318-01 (NIH)
Record Dates: First submitted 2018-07-16; First posted 2019-03-04 (Actual); Last update posted 2019-03-04 (Actual); Status verified 2019-03

CONDITIONS: Opioid Use Disorder; Substance Use Disorders; Dopamine Dysregulation Syndrome; African Americans
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders | interventions — KB220Z

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two or more groups in parallel for the duration of the study
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutraceutical, KB220Z (Experimental): A nutraceutical pill containing pro-dopamine precursors
  Interventions: Dietary Supplement: KB220Z
- Placebo (Placebo Comparator): A placebo that looks the same and is in a similar bottle
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: KB220Z — Acts to enhance dopamine
  Other Names: KB220; Synaptamine
  Arms: Nutraceutical, KB220Z
Dietary Supplement: Placebo — A placebo that looks the same, but does not contain amino acid precursors or any active ingredients in the nutraceutical
  Arms: Placebo

SUMMARY:
The investigators hypothesize that opioid use in African-Americans will be associated with hypodopaminergic alleles that alter the threshold for activating feelings of reward and pleasure within the dopaminergic system, and that these allelic frequencies will differ significantly from European Americans. Planned is a targeted system to study genetic risks for reward deficiency using risk gene panel to assign a genetic addiction risk score (GARS), comprehensive surveys to determine quality of life and exposure to stressors and trauma. This system will allow prediction of addiction and relapse potential and delivery of personalized treatment.

DETAILED DESCRIPTION:
Individuals seeking treatment for Opioid Use Disorder in the Washington DC metro area will be recruited to this Study, which consists of 1) early pre-disposition diagnosis using the Genetic Addiction Risk Score (GARS); 2) Assessment of reward deficiency, co-morbid neuropsychiatric disease, quality of life/happiness, stressors/trauma and other psychometric measurements using validated questionnaires; Urine drug testing during actual treatment that uses comprehensive analysis of reported drugs to determine compliance with prescription medications and non-abstinence to illicit drugs; and 4) adjunctive treatment with neuroadaptogen amino acid therapy (NAAT), a glutaminergic-dopaminergic optimization nutraceutical (generic name: KB220) compared to placebo, aimed to prevent relapse by induction of dopamine homeostasis.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to consent and understand questions being asked during surveys
* Must be willing to undergo pharmacogenetic testing
* Must be able to swallow tablets

Exclusion Criteria:

* Clinical Diagnosis of Alzheimer's disease/Dementia
* Clinical Diagnosis of Schizophrenia
* Clinical Diagnosis of a terminal disorder

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2018-06-16 (Actual); Primary Completion 2019-08-30 (Estimated); Study Completion 2019-08-30 (Estimated)

PRIMARY OUTCOMES:
Drug Relapse | 4 months
  Number of times opioids and other types of drugs of abuse are detected in urine
Genetic Testing for the number of risk alleles for Reward Genes through GARS | Month 1
  Number of reward gene variants in opioid use disorder patients compared to controls
Change in assessment of depression, anxiety, PTSD | 4 months
  Change from Baseline in from the Comprehensive Universal Behavioral Screen for depression, anxiety, PTSD, after 4 months
Change in Reward Deficiency Syndrome Questionnaire (RDSQ) | 4 months
  Change in risky behaviors
Addiction Severity Index (ASI) | 4 months
  Change in indices associated with addiction and associated behaviors
Vitamin B6 testing | Month 4
  Presence of B6 in blood to test for compliance with Nutraceutical

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Howard University, Washington D.C., District of Columbia
  - Medical Home Development Group, Washington D.C., District of Columbia

IPD SHARING:
Plan to Share IPD: Yes
The genetic data will be shared when compiled
Supporting Information: CSR
Time Frame: within 18 months following completion of the study, and the cleaning of clinical and genomic data